CLINICAL TRIAL: NCT02190695
Title: Leukemia SPORE Phase II Randomized Study of Decitabine Versus Decitabine and Carboplatin Versus Decitabine and Arsenic in Relapsed, Refractory, and Elderly Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Brief Title: Leukemia SPORE Phase II DAC Study for R/R and Elderly Acute AML and MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21357; NCT02188706 (obsolete NCT alias)
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Decitabine; Carboplatin; Arsenic Trioxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (3):
- Decitabine (Active Comparator): Decitabine 20mg/m2 IV over 1hour daily times 5 days every 28 days
  Interventions: Drug: Decitabine
- Decitabine and Carboplatin (Experimental): Decitabine 20mg/m2 IV over 1hour daily times 5 days, plus Carboplatin AUC 5 IV over 1hour on day 8. repeat every 28 days.
  Interventions: Drug: Decitabine; Drug: Carboplatin
- Decitabine and Arsenic (Experimental): Decitabine 20mg/m2 IV over 1 hour daily for 5 days plus Arsenic Trioxide 0.15mg/kg IV daily for 5 days. repeat every 28 days
  Interventions: Drug: Decitabine; Drug: Arsenic trioxide

INTERVENTIONS:
Drug: Decitabine — 20 mg/m2 by vein daily over 1 hour on Days 1-5 of each 28 day cycle.
  Other Names: Dacogen
Drug: Carboplatin — AUC 5 by vein over 1 hour on Day 8 of each 28 day cycle.
  Other Names: cis-Diammine; Paraplatin; Paraplatin-AQ
  Arms: Decitabine and Carboplatin
Drug: Arsenic trioxide — 0.15 mg/kg by vein over 1 hour on Days 1-5 of each 28 day cycle.
  Other Names: ATO
  Arms: Decitabine and Arsenic

SUMMARY:
The purpose of this study is to find a new way to treat Acute Myeloid Leukemia (AML), Myelodysplastic Syndrome (MDS) and Chronic Myelomonocytic Leukemia (CMML). All the drugs are used to treat AML and MDS but are not usually combined together. The investigators are looking at both the safety and Efficacy of each combination.

DETAILED DESCRIPTION:
Study Groups:

If the participant is found to be eligible to take part in this study and he/she is one of the first 30 participants enrolled, the participant will have an equal chance of being in one of 3 study groups. If the participant enrolls after the first 30 participants are enrolled, he/she will have a higher chance of being assigned to the group is having better results.

* If participant is in Group 1, he/she will receive decitabine alone.
* If participant is in Group 2, he/she will receive decitabine and carboplatin.
* If participant is in Group 3, he/she will receive decitabine and arsenic trioxide.

Study Drug Administration:

Every 4 weeks is a study cycle.

The participant will receive decitabine by vein over about 1 hours on Days 1-5 of each cycle.

If the participant is receiving carboplatin, he/she will receive it over 1 hour on Day 8 (+/-2 days) of each cycle.

If the participant is receiving arsenic trioxide, he/she will receive it over about 1 hour on Days 1-5 of each cycle

Study Visits:

Blood (about 1-2 teaspoons) will be drawn 1-2 times a week during Cycle 1 and then every 2-4 weeks after that for routine tests. If you have stable disease, blood will only be drawn every 4-6 weeks.

On Day 28 of Cycle 3 (+/- 3 days), the participant will have a bone marrow aspirate and biopsy to check the status of the disease. After that, the participant will have bone marrow biopsies/aspirations when the doctor thinks it is needed.

If the participant is in Group 3, he/she will have EKGs on Day 1 of each cycle before receiving the study drugs. On Days 1 and 4 of each cycle, blood (about 1-2 teaspoons) will also be drawn for routine tests before their dose of the study drugs.

If the participant is taken off study, blood (about 1-2 teaspoons) will be drawn for routine tests.

Length of Study:

The participant may continue taking the study drugs for as long as the doctor thinks it is in your best interest. The participant will no longer be able to take the study drug(s) if the disease gets worse, if intolerable side effects occur, or if he/she is unable to follow study directions.

This is an investigational study. Arsenic trioxide is FDA approved and commercially available for the treatment of APL. Decitabine is FDA approved and commercially available for the treatment of MDS. Carboplatin is FDA approved and commercially available for the treatment solid tumors. The study drug or study drug combination the participant receives on this study are considered investigational.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AML, relapsed or refractory to standard therapy or elderly patients with AML (age 65 or over). Patients who have AML and are younger than age 65 but considered unfit for conventional chemotherapy are eligible. Patients with de novo or treated MDS or CMML INT-1 or above are eligible. Patients may have had prior exposure to azacitidine but no more than one cycle of decitabine. Patients must have been off chemotherapy for 2 weeks prior to entering this study and have recovered from the toxicities of that therapy; A caveat to this is in the case of rapidly progressive disease. Hydroxyurea is permitted for control of elevated WBC prior to treatment and can be continued for the first 4 weeks of therapy. Erythropoiesis stimulating agents (ESAs) and GCSF are allowed before therapy. ESAs, GCSF or other growth factors are permitted on therapy.
2. Performance 0-2 (ECOG).
3. Adequate cardiac functions assessed by 2D ECHO (NYHA cardiac III-IV excluded).
4. Pre-treatment EKG
5. Adequate end organ function with creatinine </= 2mg/dL and total bilirubin </= 2mg/dL, AST and ALT </= or = 2.5 X institutional ULN.
6. Absence of significant intercurrent illness such as uncontrolled heart failure, unstable angina, cardiac arrhythmia and psychiatric illness which precludes the giving of informed consent.
7. Signed informed consent

Exclusion Criteria:

1. Nursing and pregnant females. Patients of childbearing potential should practice effective methods of contraception. Should a woman become preg-nant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
2. Current uncontrolled infections.
3. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Chronic kidney disease > stage 3.
5. HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Time to complete or partial remission | up to 16 weeks
  evaluation of the complete and partial response rates (antileukemic effect) and the amount of time taken to achieve the response.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Kropf, MD, Principal Investigator — Temple University Health System
Locations (2):
- United States (2):
  - Temple BMT Program at Jeanes Hospital, Philadelphia, Pennsylvania
  - M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Kropf PL, Chung W, Shameem R, Xiao L, Balch C, Huang X, Issa JJ. A phase 2 study of decitabine with or without carboplatin and arsenic trioxide in patients with MDS and AML. Blood Neoplasia. 2025 Jan 23;2(2):100071. doi: 10.1016/j.bneo.2025.100071. eCollection 2025 May. PMID 40453133